CLINICAL TRIAL: NCT04062695
Title: Efficacy of Tofacitinib in Reduction of Inflammation Detected on MRI in Patients With Psoriatic ArthritiS PresenTing With Axial InvOlvement - a Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial
Brief Title: Tofacitinib for Reduction of Spinal Inflammation in Patients With Psoriatic ArthritiS PresenTing With Axial InvOlvement
Acronym: PASTOR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Denis Poddubnyy, Prof. Dr. Denis Poddubnyy, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PASTOR2018
Record Dates: First submitted 2019-05-14; First posted 2019-08-20 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Psoriatic Arthritis; Spondylitis; Sacroilitis
Keywords: Psoriatic Arthritis; Sacroiliitis; Spondylitis; MRI
MeSH Terms: conditions — Arthritis, Psoriatic; Spondylitis; Sacroiliitis | interventions — tofacitinib; Tablets

STUDY DESIGN:
Intervention Model Description: Placebo controlled parallel group for 12 weeks followed by 12 weeks open label
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tofacitinib (Active Comparator): 5 mg oral BID
  Interventions: Drug: Tofacitinib 5 MG Oral Tablet [Xeljanz]
- Placebo (Placebo Comparator): matching Placebo BID
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Tofacitinib 5 MG Oral Tablet [Xeljanz] — verum tablets
  Other Names: Xeljanz
  Arms: Tofacitinib
Drug: Placebo oral tablet — tablets containing placebo
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of Tofacitinib in reducing inflammation in the sacroiliac joints and spine on magnetic resonance imaging (MRI) in patients with active Psoriatic Arthritis (PsA) with axial Involvement (BASDAI [Bath Ankylosing Spondylitis Disease Activity Index] ≥ 4 and total backpain ≥ 4 despite treatment with NSAIDs plus evidence of active inflammation in the sacroiliac joints or spine on MRI).

DETAILED DESCRIPTION:
This study is a prospective, randomized, double-blind, placebo-controlled, multicenter study to investigate the efficacy of Tofacitinib in reducing inflammation in the sacroiliac joints and in the spine on MRI in patients with active axial PsA.

Eligible patients (n=80) will be randomized 1:1 to receive either Tofacitinib 5mg orally twice daily or placebo for a 12-week period. After week 12, all patients will receive Tofacitinib 5mg orally twice daily for another 12 weeks. The study duration will include a 6-week screening period, a 24-week treatment period and a safety follow-up period of 4 weeks. Patients will be closely monitored throughout the study on a total of 11 visits. Safety data will be collected in the form of adverse events, vital parameters, physical examinations, and laboratory parameters throughout the study.

The baseline MRI of the whole spine and sacroiliac (SI) joints will be performed within the 6-week screening period to confirm the presence of active inflammation (bone marrow edema) compatible with Spondyloarthritis (will be assessed by a central reader), at week 12 to evaluate the primary study endpoint, and at week 24 to evaluate the secondary endpoint.

The primary study endpoint will be an improvement of the total Berlin MRI score for sacroiliac joints and spine at week 12 as compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Psoriatic Arthritis fulfilling ClASsification for Psoriatic ARthritis (CASPAR) criteria
* chronic back pain > 3 months
* BASDAI value ≥ 4 and backpain ≥ 4 / 10 VAS
* presence of active inflammation in Screening MRI of sacroiliac joints and / or spine (central reading)
* history of inadequate response to ≥ 2 NSAIDs or intolerance / contraindications

Exclusion Criteria:

* active current infection, severe infections in the last 3 months
* history of recurrent Herpes zoster or disseminated Herpes simplex
* immunodeficiency
* chronic Hepatitis B, C or HIV infection
* women: pregnant or lactating (have to practice reliable method of contraception)
* other severe diseases conflicting with a clinical study, contraindications for MRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-08-04 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
MRI Berlin Score | Week 12 vs Baseline
  Improvement of the Berlin MRI score for sacroiliac joints and spine. Scoring includes spinal inflammation (Lucas C et al, J Rheumatol 2007): 23 vertebral units with semiquantitative range of inflammation between 0 to 3 (min. score = 0, max. score = 69, the higher the worse). Additionally, inflammation of the sacroiliac joints is scored (Hermann KG, Rheumatologe 2004; scoring each quadrant between 0 and 4, max. score 16, the higher, the worse).

SECONDARY OUTCOMES:
The Assessment of Spondyloarthritis International Society (ASAS) response criteria | Week 12 vs Baseline, Week 24 vs Baseline, Week 24 vs Week 12
  Assessment of Spondyloarthritis International Society Response Criteria (Anderson JJ, Arthritis Rheum 2001): change in percent of at least 3 of 4 subcores (Patient Global VAS, Pain VAS, BASFI and BASDAI questions 5&6).
Responses in ASAS Health Index | Week 12 vs Baseline, Week 24 vs Baseline, Week 24 vs Week 12
  Assessment of Spondyloarthritis International Society ASAS Health Index (Kiltz U, Ann Rheum Dis 2015). Consisting of 17 questions answered, calculated in percent (100 % = best spondylarthritis related health).
Responses in ASDAS | Week 12 vs Baseline, Week 24 vs Baseline, Week 24 vs Week 12
  Ankylosing Spondylitis Disease Activity Score (ASDAS) combining 3 questions VAS (back pain, peripheral pain and morning stiffness) with CRP or ESR; formulas used as described in Lucas C, Ann Rheum Dis 2009. Values <1.3 inactive disease, <2.1 low disease activity, 2.1-3.5 high disease activity, >3.5 very high disease activity.
Responses in BASDAI | Week 12 vs Baseline, Week 24 vs Baseline, Week 24 vs Week 12
  Bath Ankylosing Spondylitis Disease Activity Index (BASDAI). Calculated score from 6 questions VAS; range 0-10, the higher the worse.
Responses in BASFI | Week 12 vs Baseline, Week 24 vs Baseline, Week 24 vs Week 12
  Bath Ankylosing Spondylitis Functional Index (BASFI). Mean of 10 questions VAS, range 0-10; higher value = more impaired function.
Responses in BASMI(lin) | Week 12 vs Baseline, Week 24 vs Baseline, Week 24 vs Week 12
  Bath Ankylosing Spondylitis Metrology Index - linear score (BASMI; van der Heijde Ann Rheum Dis 2008). Measuring Schober´s test (cm), intermalleolar distance (cm), cervical rotation (degree), lateral lumbar flexion (cm) and tragus-to-wall-distance (cm) and calculate the score as reported in the citation.
Responses in HAQ-DI | Week 12 vs Baseline, Week 24 vs Baseline, Week 24 vs Week 12
  Health assessment questionnaire disability index (HAQ-DI; Princus T, Arthritis Rheum 1983) measuring influence of arthritis on quality of life. Patient questionnaire recalculated in scores 0 to 3, higher = worse.
Responses in Patient Global Score | Week 12 vs Baseline, Week 24 vs Baseline, Week 24 vs Week 12
  Patient Global Score of overall disease activity - VAS 0-10 (higher = worse)
Responses in Physician Global Score | Week 12 vs Baseline, Week 24 vs Baseline, Week 24 vs Week 12
  Physician Global Score of overall disease activity - VAS 0-10 (higher = worse).
Responses in DAPSA | Week 12 vs Baseline, Week 24 vs Baseline, Week 24 vs Week 12
  Disease Activity in PSoriatic Arthritis (DAPSA; Schoels M, Arthritis Rheum 2010); calculated by summing swollen joint count (max. 66) + tender joint count (max. 68) + patient pain VAS + patient global assessments VAS + CRP. Value ranges 0 to >28 (the higher, the worse).
Responses in PASI | Week 12 vs Baseline, Week 24 vs Baseline, Week 24 vs Week 12
  Psoriasis Area and Severity Index (PASI) - description of skin involvement regarding scaling, redness, thickness and body surface area. Range 0-72.
Responses in MASES | Week 12 vs Baseline, Week 24 vs Baseline, Week 24 vs Week 12
  Maastricht Ankylosing Spondylitis Enthesitis Score (MASES;Heuft-Dorenbosch Ann Rheum Dis 2003). Assessing 13 clinical enthesial sites (yes / no). Range 0-13.
Response in CRP | Week 12 vs Baseline, Week 24 vs Baseline, Week 24 vs Week 12
  C-reactive protein (CRP, mg per litre)
Response in ESR | Week 12 vs Baseline, Week 24 vs Baseline, Week 24 vs Week 12
  Erythrocyte Sedimentation Rate (ESR, mm per 1 hour)
MRI Berlin Score | Week 24 vs Baseline, Week 24 vs Week 12
  Improvement of the Berlin MRI score (description see primary outcome) for sacroiliac joints and spine

CONTACTS AND LOCATIONS:
Overall Officials: Denis Poddubnyy, Prof, Principal Investigator — Charite University, Dept. Rheumatology CBF
Locations (19):
- Germany (19):
  - Charite University, Rheumatology CCM, Berlin
  - Praxis für Rheumatologie, Berlin
  - Charite University - Dept. Rheumatology CBF, Berlin
  - University Cologne, Dept. Rheumatology, Cologne
  - Uniklinik, Forschungszentrum Rheumatologie, Düsseldorf
  - Praxis Dilltal, Ehringshausen
  - Uniklinikum, Med. Klinik 3, Erlangen
  - CIRI Zentrum f innovative Diagnsotik und Therapie, Frankfurt am Main
  - Uniklinikum, Dept. Rheumatologie, Freiburg im Breisgau
  - Hamburger Rheumaforschungszentrum, Hamburg
  - Rheumazentrum Ruhrgebiet, Herne
  - Uniklinik, Rheumatologie, Kiel
  - Klinikum Ludwigshafen, Rheumatologie, Ludwigshafen
  - Rheumapraxis Dr. Sieburg, Magdeburg
  - Inst. f Präventive Medizin & Klinische Forschung, Magdeburg
  - Uniklinikum, I. Med. Klinik, Mainz
  - Praxis Prof. Kellner, München
  - Rheumatol Schwerpunktpraxis, Steglitz
  - KH St. Josef, Dept. Rheumatology, Wuppertal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Proft F, Torgutalp M, Muche B, Rios Rodriguez V, Verba M, Poddubnyy D. Efficacy of tofacitinib in reduction of inflammation detected on MRI in patients with Psoriatic ArthritiS presenTing with axial involvement (PASTOR): protocol of a randomised, double-blind, placebo-controlled, multicentre trial. BMJ Open. 2021 Nov 16;11(11):e048647. doi: 10.1136/bmjopen-2021-048647. PMID 34785545